CLINICAL TRIAL: NCT00505596
Title: Expanded Prenatal Testing Options and Informed Choice
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); March of Dimes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01HD049686 (NIH); R01HD049686 (NIH); 12-FY09-213 (Other Grant/Funding Number: March of Dimes)
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Pregnancy Related
Keywords: Prenatal testing; Decisionmaking; Decision aid; Informed choice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized decision aid (Experimental): Participants instructed to view the updated PT Tool and told that they can have whatever tests they would like (including no tests) and that tests that are not covered by their insurance will be paid for by the study (Informed free choice). They also participate in a baseline pre-randomization interview and one follow-up telephone interview.
  Interventions: Behavioral: Informed free choice
- Usual care (No Intervention): Control group, in which participants receive no intervention beyond a baseline pre-randomization interview and one follow-up telephone interview.

INTERVENTIONS:
Behavioral: Informed free choice — Women will be instructed to view an updated prenatal testing decision aid and will be told that they can have whatever tests they would like (including no tests) and that tests that are not covered by their insurance will be paid for by the study
  Arms: Computerized decision aid

SUMMARY:
The proposed study will determine the impact of providing complete information about all prenatal tests for chromosomal disorders to racially/ethnically and sociodemographically diverse women of all ages and allowing them to make informed choices regarding which tests - if any - to undergo. Specifically, we propose to update a validated prenatal testing decision-assisting tool ("PT Tool") to incorporate new screening options and make it more accessible to lower literacy and culturally diverse populations. We then will conduct a randomized controlled trial comparing the effect of an "informed free choice" approach consisting of providing complete information regarding and access to all prenatal testing options to that of usual care among a diverse population of pregnant women.

DETAILED DESCRIPTION:
Our primary goal is to generate evidence needed to determine whether clinicians should consider an alternative to the current practice of using risk-based thresholds for invasive testing that would allow all women to make informed choices reflective of their values and preferences. A second goal is to expand PT Tool to include new screening tests and modify it for clinical use by lower literacy populations, so that pregnant women of diverse backgrounds will have accurate and unbiased information about the complex array of testing options, thereby minimizing barriers to and disparities in informed choice.

Specific Aim 1) Determine which testing strategies are selected by a racially/ethnically, socioeconomically, and age-diverse group of pregnant women who receive complete information on all testing options and have all options available to them compared to women receiving usual care.

Specific Aim 2) Update the English-language version of PT Tool and create a Spanish-language version to include the most up-to-date information on new and forthcoming prenatal screening options and modify it for use in clinics by women of varying literacy levels.

Specific Aim 3) Assess the impact of receiving complete information on all testing options and having all options available on knowledge, risk comprehension, and decisional conflict compared to usual care.

We will perform an open, parallel-comparison randomized clinical trial of an "informed free choice" approach to prenatal testing to usual care in 1200 women presenting for prenatal care by 20 gestational weeks. 600 women will be randomized to usual care, the control group, in which they will receive no intervention beyond a baseline pre-randomization interview and a follow-up telephone interview. The other 600 women will be randomized to "informed free choice," in which they will be instructed to view the updated PT Tool and will be told that they can have whatever tests they would like (including no tests) and that tests that are not covered by their insurance will be paid for by the study. They also will participate in a follow-up telephone interview.

Revised clinicaltrials.gov protocol. The original study design was proposed and funded during the era when guidelines from the American College of Obstetricians and Gynecologists (ACOG) regarding access to prenatal testing differed by maternal age stratum (less than 35 years at the age of delivery versus 35 years or older). Our original primary hypothesis posited that the effect of IFC would increase invasive test use among women who were less than 35 years old while decreasing invasive test use among women 35 years or older. The thought underlying this hypothesis was that the younger women, who traditionally were not informed of this option, and for whom insurance coverage for these procedures was not consistently available, would increase their overall invasive test use if these informational and financial barriers to were removed in the context of the study. On the other hand, women 35 years and older, for whom the offer of invasive diagnostic testing was considered routine, would become more informed about the risks and benefits of both screening and invasive diagnostic testing, would be less likely to default to invasive testing. The original sample size estimate was N=1200 women.

After we began enrolling women in the study and the new ACOG guidelines were issued, the prenatal testing decision support guide we had created was out-of-date with respect to the array of available prenatal screening and diagnostic tests and restrictions on invasive test use based upon maternal age. We therefore decided to end the original trial (N=381). We completely revised the decision support guide to describe the new screening options and better represent the current policy landscape. We also reformulated our primary hypothesis to eliminate the age dichotomy, and initiated a new randomized trial using the revised decision support guide to be completed within the time and budgetary constraints of the initially funded project.

Our primary hypothesis was that women who were randomized to informed free choice would undergo invasive prenatal diagnostic testing at a lower rate than women randomized to the usual care group, regardless of maternal age. Given that the restrictions on access to testing based upon maternal age had been eliminated, we hypothesized that women of all ages who were randomized to informed free choice would have lower invasive test use rates compared to women randomized to usual care. In our study of trends in the use of invasive diagnostic testing among women who delivered at an integrated health care system in California, we found that the number of amniocenteses and CVS procedures performed as a percentage of the total number of deliveries in 2006 was 12.1% (Norton ref). Assuming N=1200-381=819 participants for the new trial, 80% power, two-tailed alpha equal to 0.05, 90% retention at follow-up, and a 12.1% invasive test use rate within the usual care group, the design was capable of detecting a group difference corresponding to an invasive test use rate of ≤6.2% in the informed free choice group (OR=2.10, a 'small-medium' effect size). We also hypothesized that compared to usual care, women in informed free choice would have increased testing knowledge and risk comprehension as well as reduced decisional conflict, regret, and pregnancy worry; the design was capable of a minimum detectable a group difference equal to d=0.21 standard deviations, which is considered a 'small' effect size.

ELIGIBILITY:
Inclusion Criteria:

* No more than 20 weeks pregnant.

Exclusion Criteria:

* Inability to speak English or Spanish.
* Those carrying triplets or higher order gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 744 (Actual)
Dates: Start 2007-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Prenatal test use | 9 months
  Information on prenatal test use was obtained from medical charts and used to classify women according to the testing strategy they underwent: no screening or diagnostic testing for chromosomal problems; starting with a screening test prior to deciding about diagnostic testing; and going straight to invasive diagnostic testing.

SECONDARY OUTCOMES:
Patient reported outcome questionnaire | 9 months
  Knowledge, risk comprehension, decisional conflict/decision regret as assessed during a 20-minute follow-up telephone interview: 5-item measure adapted from the Maternal Serum Screening Knowledge Questionnaire; risk comprehension was assessed by asking participants to estimate, out of 1000 pregnant women who had an amniocentesis, how many would experience a miscarriage caused by the procedure (women who reported the risk to be greater than zero but less than 10 were scored as correct), and out of 1000 pregnant women their age, how many are carrying a fetus affected by Down syndrome (we compared this risk to the participant's age-related Down syndrome risk and scored concordant replies as correct); decisional conflict and regret were assessed using 15-items from the Decisional Conflict Scale and the 5-item Decision Regret Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kuppermann, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Kuppermann M, Pena S, Bishop JT, Nakagawa S, Gregorich SE, Sit A, Vargas J, Caughey AB, Sykes S, Pierce L, Norton ME. Effect of enhanced information, values clarification, and removal of financial barriers on use of prenatal genetic testing: a randomized clinical trial. JAMA. 2014 Sep 24;312(12):1210-7. doi: 10.1001/jama.2014.11479. PMID 25247517